CLINICAL TRIAL: NCT04158219
Title: Development of an Integrated Depression and Behavioral Risk Factor Reduction Intervention for Secondary Prevention Following Acute Coronary Syndrome
Brief Title: Healthy Heart Habits
Acronym: H^3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Andrew Busch, Sr. Clinical Psychologist, Associate Professor, Hennepin Healthcare Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R03HL136540 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome; Depression
Keywords: Behavioral randomized control trial; Behavioral activation; Multiple health behavior change; Integrated care
MeSH Terms: conditions — Acute Coronary Syndrome; Depression | interventions — Health

STUDY DESIGN:
Intervention Model Description: Twenty subjects will be given the intervention according to the treatment manual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Behavioral activation for health and depression (BA-HD)
  Interventions: Behavioral: Behavioral activation for health and depression (BA-HD)

INTERVENTIONS:
Behavioral: Behavioral activation for health and depression (BA-HD) — Consistent with successful BA manuals, we plan to conduct up to 10 sessions of treatment over 12 weeks (the recommendation will be at least 8 sessions; scheduling of sessions will be flexible and conform to patient preference). The initial two sessions will be about 50 minutes long and later sessions will be 20-30 minutes long. Sessions can be done on site or over the phone; home visits will be offered for sessions 1-2 if a participant cannot travel. Treatment sessions will use behavioral activation techniques to assess participant values and link these values to behavior change. Goal-setting will focus on sequential, idiographic behavior change (tobacco use, medication adherence, physical activity, and diet) and be accompanied by educational materials and commercially available tools (e.g. activity trackers, pillboxes).

SUMMARY:
Approximately 350,000 Acute Coronary Syndrome (ACS) patients experience significant depression symptoms each year in the US. Post-ACS depressed mood interferes with patients making necessary changes to behavioral risk factors (e.g., smoking cessation) and predicts poor medical outcomes. The proposed study will develop an integrated depression and behavioral risk factor reduction intervention for secondary prevention post-ACS through an open trial of 20 patients.

DETAILED DESCRIPTION:
Depression predicts high rates of morbidity/mortality among acute coronary syndrome (ACS) patients. Part of this relationship is explained by a poor profile of behavioral risk factors (i.e., smoking,physical activity, medication adherence, diet). An integrated treatment targeting both depressed mood and multiple behavioral risk factors could be highly effective in reducing post-ACS mortality. Behavioral Activation for depression may be an ideal counseling treatment for this since it has recently shown promise for facilitating behavioral risk factor changes in ACS patients with depression (K23HL107391). The current study adapts this manual targeting post-ACS depressed mood and smoking cessation to target depression and multiple behavioral risk factors post-ACS. This study will be an open trial (N=20) to test the feasibility and acceptability of our procedures and obtain initial indications of efficacy. This study hypothesizes that 1) the BA-HD manual and study procedures will be feasible and acceptable to post-ACS patients with depressed mood as measured by self-report, recruitment/retention rate, and post- treatment qualitative interviews and 2) that participants will experience clinically significant improvements in depressed mood and behavioral risk factor profile. The long-term goal of this research is to improve long-term survival rates following ACS.

ELIGIBILITY:
Inclusion criteria:

* ACS diagnosis (diagnosis of unstable angina, ST and non-ST elevation myocardial infarction) documented in medical record in the preceding 2-12 months
* Current diagnosis of depression documented in medical record, OR clinically administered PHQ-9 score of 10 or greater documented in the medical record in the preceding 12 months, OR CES-D score greater than or equal to 10
* current non-adherence to 1 or more of 4 more behavioral risk factors
* willing to make immediate changes to one or more of the relevant behavioral risk factors
* age of 18-75
* lives within 1.5 hours of Hennepin Healthcare
* fluent in English.

Exclusion criteria:

* Limited mental competency (as indicated in medical chart)
* presence of current exacerbation of psychosis/serious mental illness or suicidality
* in hospice care
* currently attending regular counseling targeting depression or any health behavior change
* currently attending a cardiac rehabilitation program (those excluded for being in rehabilitation will be re-contacted after completion)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Busch, PhD, Principal Investigator — Hennepin Healthcare
Locations (1):
- Hennepin Healthcare, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gathright EC, Vickery KD, Ayenew W, Whited MC, Adkins-Hempel M, Chrastek M, Carter JK, Rosen RK, Wu WC, Busch AM. The development and pilot testing of a behavioral activation-based treatment for depressed mood and multiple health behavior change in patients with recent acute coronary syndrome. PLoS One. 2022 Feb 3;17(2):e0261490. doi: 10.1371/journal.pone.0261490. eCollection 2022. PMID 35113860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 8
Completed | 7
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.88 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Acceptability Measured by the Client Satisfaction Questionnaire
Description: This will be assessed at the end of the intervention using the 8-item Client Satisfaction Questionnaire. score range 8-32 with higher score indicating greater satisfaction.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 7
score on a scale | 30.57 (2.23)

2. Primary Outcome: Treatment Engagement Measured by Sessions Attended
Description: Throughout the study we will measure engagement by tracking attendance of treatment sessions.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: sessions attended
Arm/Group | Treatment
Number analyzed (Participants) | 7
sessions attended | 8.65 (2.77)

3. Secondary Outcome: Study Retention Measured by the Number of Participants Who Complete the Follow-up Assessments
Description: Study retention will be tracked by measuring the number of participants who complete the follow-up assessments
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 8
Participants | 7

4. Secondary Outcome: Depression Symptoms as Measured by PHQ-9 (Patient Health Questionnaire-9)
Description: Depression symptoms will be measured by Patient Health Questionnaire, 9-item.Score range is 0-27 with higher scores indicating higher depression symptoms.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 7
score on a scale
  Baseline | 8.29 (5.12)
  12 Weeks | 4.86 (3.89)

5. Secondary Outcome: Depression Symptoms as Measured by CES-D 10 (Center for Epidemiological Studies Depression Scale Revised)
Description: Depression symptoms will also be measured by the Center for Epidemiological Studies Depression scale 10-item. Score range is 0-30 with higher scores indicating higher depression symptoms.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 7
score on a scale
  Baseline | 11.43 (4.72)
  12 Weeks | 8.57 (4.54)

6. Secondary Outcome: Composite Behavioral Risk Factor Adherence MOS (Medical Outcomes Study Patient Adherence Questionnaire)
Description: The Medical Outcomes Study Patient Adherence Questionnaire will be used to assess adherence to behavior change goals.10 items related to cardiac health will be scored. Items are rated on a 1-6 scale. Because not all items will be relevant to all participants, the average score across the relevant items for each participant will be presented. Higher scores indicating greater adherence to healthcare provider recommendations.
Time Frame: At 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 7
score on a scale
  Baseline | 3.75 (.94)
  12 weeks | 4.53 (.70)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT04158219/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT04158219/SAP_001.pdf
  • Informed Consent Form (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT04158219/ICF_002.pdf